CLINICAL TRIAL: NCT07090746
Title: Evaluation of Dentoalveolar Changes of Clear Aligners Versus Fixed Orthodontic Appliances on Skeletal Class I Non-extraction Patients With Dental Crowding: Randomized Controlled Clinical Trial
Brief Title: Evaluation of Dentoalveolar Changes of Clear Aligners Versus Fixed Orthodontic Appliances on Skeletal Class I Non-extraction Patients With Dental Crowding
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Kholod Elbady, Assistant lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A0208023OR
Record Dates: First submitted 2025-06-02; First posted 2025-07-29 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-07

CONDITIONS: Skeletal Class I Non-extraction Patients With Dental Crowding
Keywords: clear aligners
MeSH Terms: interventions — Orthodontic Appliances, Removable; Orthodontic Appliances, Fixed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non extraction crowding cases for clear aligner (Active Comparator)
  Interventions: Device: Clear aligner
- Non extraction crowding cases for fixed orthodontic appliance (Active Comparator)
  Interventions: Device: Fixed orthodontic appliance

INTERVENTIONS:
Device: Clear aligner — Clear aligner
  Arms: Non extraction crowding cases for clear aligner
Device: Fixed orthodontic appliance — Fixed orthodontic appliance
  Arms: Non extraction crowding cases for fixed orthodontic appliance

SUMMARY:
To evaluate dentoalveolar changes of clear aligners versus fixed orthodontic appliances on skeletal class I non-extraction patients with dental crowding.

ELIGIBILITY:
Inclusion Criteria:

* Complete permanent dentition.
* Angle Class I malocclusion cases with mild to moderate crowding (2-6 mm) that can be resolved by dental expansion and interproximal reduction (IPR).
* Good oral hygiene.

Exclusion Criteria:

* Bad oral hygiene.
* Previous orthodontic treatment.
* Periodontal disease and previous periodontal surgery procedures.
* Systemic diseases and/or craniofacial syndromes.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Alveolar bone thickness | From date of randomization until the date of first documented acceptable teeth alignment, assessed up to 12 months.
  Alveolar bone thickness will be assessed in vestibular and oral sides, parallel to the cervical reference line (CRL) at 3 different evels and expressed in millimeters.
Alveolar bone height | From date of randomization until the date of first documented acceptable teeth alignment, assessed up to 12 months.
  Alveolar bone height loss will be measured perpendicularly to the CRL in both vestibular and oral sides. It will be represented as the difference between pretreatment and post treatment distance from alveolar crest to the CRL, expressed in millimeters.

SECONDARY OUTCOMES:
Comparison of transverse dental changes between the two groups. | From date of randomization until the date of first documented acceptable teeth alignment, assessed up to 12 months.
  Assessment of inter-molar and inter-canine widths
Assessment of Apical root resorption | From date of randomization until the date of first documented acceptable teeth alignment, assessed up to 12 months.
  comparison of root length changes after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided